CLINICAL TRIAL: NCT01247571
Title: A Phase II Evaluation of Pazopanib (NSC # 737754) in the Treatment of Recurrent or Persistent Carcinosarcoma of the Uterus
Brief Title: Pazopanib Hydrochloride in Treating Patients With Recurrent or Persistent Uterine Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02658; NCI-2011-02658 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0230D; CDR0000689585; GOG-0230D (Other: NRG Oncology); GOG-0230D (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Results first posted 2017-07-27 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Recurrent Uterine Corpus Sarcoma; Uterine Carcinosarcoma
MeSH Terms: interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pazopanib hydrochloride) (Experimental): Patients receive pazopanib hydrochloride PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pazopanib Hydrochloride

INTERVENTIONS:
Drug: Pazopanib Hydrochloride — Given PO
  Other Names: GW786034B; Votrient

SUMMARY:
This phase II trial studies how well pazopanib hydrochloride works in treating patients with uterine cancer that has come back or has not responded to treatment. Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Pazopanib hydrochloride may also stop the growth of uterine cancer by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the activity of pazopanib in patients with persistent or recurrent carcinosarcoma of the uterus as measured by the proportion of patients who survive progression-free for at least 6 months and the proportion of patients who have objective tumor response (complete or partial).

SECONDARY OBJECTIVES:

I. To determine the frequency and severity of adverse events as assessed by Common Terminology Criteria of Adverse Events version 4.0 (CTCAE v4.0).

II. To determine the duration of progression-free survival and overall survival.

OUTLINE: This is a multicenter study.

Patients receive pazopanib hydrochloride orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed uterine carcinosarcoma which is persistent or recurrent; acceptable histological type is defined as carcinosarcoma (malignant mixed müllerian tumor), homologous or heterologous type
* Patients must have measurable disease

  * Measurable disease is defined by Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1)
  * Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded)
  * Each lesion must be greater than or equal to 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI), or caliper measurement by clinical exam or greater than or equal to 20 mm when measured by chest x-ray
  * Lymph nodes must be greater than or equal to 15 mm in short axis when measured by CT or MRI
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST version 1.1

  * Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must not be eligible for a higher priority Gynecologic Oncology Group (GOG) protocol, if one exists

  * In general, this would refer to any active GOG phase III protocol or rare tumor protocol for the same patient population
* Patients must have a GOG performance status of 0, 1, or 2
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy

  * Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
  * Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration
  * Any other prior therapy (chemotherapy) directed at the malignant tumor, must be discontinued at least three weeks prior to registration
  * At least 4 weeks must have elapsed since the patient underwent any major surgery (e.g., major: hysterectomy, resection of a lung nodule - minor: central venous access catheter placement)
* Patients must have had one prior chemotherapeutic regimen for management of carcinosarcoma; initial treatment may include chemotherapy, chemotherapy and radiation therapy, and/or consolidation/maintenance therapy; chemotherapy administered in conjunction with primary radiation as a radio-sensitizer WILL be counted as a systemic chemotherapy regimen
* Patients are allowed to receive, but are not required to receive, one additional cytotoxic regimen for management of recurrent or persistent disease according to the following definition:

  * Cytotoxic regimens include any agent that targets the genetic and/or mitotic apparatus of dividing cells, resulting in dose-limiting toxicity to the bone marrow and/or gastrointestinal mucosa
  * Note: patients on this non-cytotoxic study are allowed to receive one additional cytotoxic chemotherapy regimen for management of recurrent or persistent disease, as defined above; however, due to the novel nature of biologic compounds, patients are encouraged to enroll on second-line non-cytotoxic studies prior to receiving additional cytotoxic therapy
  * Patients must have NOT received any non-cytotoxic chemotherapy for management of recurrent or persistent disease; prior hormonal therapy is permitted
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcL
* Platelets greater than or equal to 100,000/mcL
* Hemoglobin level greater than or equal to 9 g/dL
* Creatinine less than or equal to 1.5 x institutional upper limit of normal (ULN)
* Urine protein/creatinine ratio (UPCR) must be less than 1 (or urinary protein less than 1.0 g/24 hours)
* Bilirubin less than or equal to 1.5 x ULN (subjects with Gilbert syndrome and elevations of indirect bilirubin only are eligible)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 2.5 x ULN
* Alkaline phosphatase less than or equal to 2.5 x ULN
* Subjects who have BOTH bilirubin greater than ULN and AST/ALT greater than ULN are not eligible

  * Specifically, if bilirubin is greater than 1 x ULN but less than or equal to 1.5 x ULN, THEN the AST and ALT must be less than or equal to ULN for patient to be eligible; if AST and/or ALT are greater than 1 x ULN but less than or equal to 2.5 x ULN, THEN the bilirubin must be less than or equal to ULN for patient to be eligible
* Prothrombin time (PT) such that international normalized ratio (INR) is less than or equal to 1.5 x ULN (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin) and a partial thromboplastin time (PTT) less than or equal to 1.5 x ULN
* Patients with a history of hypothyroidism/hyperthyroidism must have had stable well-controlled thyroid function for a minimum of 2 months as a condition for eligibility and that all other patients must have normal baseline thyroid function tests (thyroid stimulating hormone [TSH], triiodothyronine [T]3, T4)
* Patients must have the ability to understand and sign an approved informed consent and authorization permitting release of personal health information
* Patients who have met the pre-entry requirements
* Patients must be capable of taking and absorbing oral medications; a patient must be clear of the following:

  * Any lesion, whether induced by tumor, radiation or other conditions, which makes it difficult to swallow tablets
  * Prior surgical procedures affecting absorption including, but not limited to major resection of stomach or small bowel
  * Active peptic ulcer disease
  * Malabsorption syndrome
* Patients must be capable of taking and absorbing oral medications
* A patient must be clear of the following:

  * Any lesion, whether induced by tumor, radiation, or other conditions, which makes it difficult to swallow tablets
  * Prior surgical procedures affecting absorption including, but not limited to, major resection of stomach or small bowel
  * Active peptic ulcer disease
  * Malabsorption syndrome
* Any concomitant medications that are associated with a risk of corrected QC (QTc) prolongation and/or Torsades de pointes should be discontinued or replaced with drugs that do not carry these risks, if possible; patients who must take medication with a risk of possible risk of Torsades de pointes should be watched carefully for symptoms of QTc prolongation, such as syncope

  * Patients with personal or family history of congenital long QTc syndrome are NOT eligible
* Strong inhibitors of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) are prohibited; grapefruit juice is also an inhibitor of CYP450 and should not be taken with pazopanib; CYP3A4 Inducers: strong inducers of CYP3A4 are prohibited; cytochrome P450 (CYP) substrates: concomitant use of agents with narrow therapeutic windows that are metabolized by CYP3A4, cytochrome P450, family 2, subfamily D, polypeptide 6 (CYP2D6), or cytochrome P450, family 2, subfamily C, poly peptide 8 (CYP2C8) is not recommended
* Patients of childbearing potential must have a negative pregnancy test prior to the study treatment and agree to be practicing an effective form of contraception throughout study treatment; pregnant women are excluded from this study

Exclusion Criteria:

* Patients who have had prior therapy with pazopanib
* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of uterine carcinosarcoma within the last three years are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of uterine carcinosarcoma within the last three years are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients with clinically significant cardiovascular disease; this includes:

  * Patients must have blood pressure (BP) no greater than 140 mmHg (systolic) and 90 mmHg (diastolic) for eligibility
  * Myocardial infarction or unstable angina within 6 months of the first date of pazopanib therapy
  * New York Heart Association (NYHA) class II or greater congestive heart failure
  * History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation) or cardiac arrhythmias requiring anti-arrhythmic medications; this does not include asymptomatic, atrial fibrillation with controlled ventricular rate
  * Women who have received prior anthracycline (e.g., doxorubicin and/or liposomal doxorubicin) and who have an ejection fraction less than the institutional lower limit of normal will be excluded from the study; patients with a prior life time exposure to doxorubicin (or liposomal doxorubicin) of greater than 300 mg/m^2 are NOT eligible
  * CTCAE grade 2 or greater peripheral vascular disease
  * History of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of pazopanib therapy
  * Women with a baseline QTc >= 480 milliseconds
  * History of cardiac angioplasty or stenting within 6 months prior to registration; history of coronary artery bypass graft surgery within 6 months prior to registration
  * A patient with arterial thrombosis within 6 months prior to enrollment
* Patients with history or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, seizures not controlled with standard medical therapy or any brain metastases
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels
* Patients with serious, non-healing wound, ulcer, or bone fracture; this includes history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days prior to the first date of pazopanib therapy; patients with underlying lesions that caused the fistula or perforation in the past that have not been corrected
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pazopanib
* Human immunodeficiency virus (HIV)-positive subjects on combination antiretroviral therapy are ineligible
* Patients who are nursing; patients who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug
* Patients with any condition that may increase the risk of gastrointestinal bleeding or gastrointestinal perforation, including:

  * Active peptic ulcer disease
  * Known gastrointestinal intraluminal metastatic lesions (gastrointestinal serosa metastatic lesion are permitted)
  * Inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease)
* History of hemoptysis in excess of 2.5 mL (1/2 teaspoon) within 8 weeks prior to first dose of pazopanib
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susana Campos, Principal Investigator — NRG Oncology
Locations (41):
- United States (41):
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Hospital Orlando, Orlando, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Sudarshan K Sharma MD Limted-Gynecologic Oncology, Hinsdale, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Oncology Center, Indianapolis, Indiana
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium CCOP, Ann Arbor, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Groups:
- Pazopanib: Pazopanib 800mg daily until disease progression or adverse effects prohibit further therapy (one cycle equals 28 days)
Period: Overall Study
Arm/Group | Pazopanib
Started | 22
Completed | 19
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Pazopanib
Number analyzed (Participants) | 19
Age, Customized [Number; unit: participants]
  50-59 | 1
  60-69 | 11
  70-79 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response (Complete or Partial)
Description: Complete and Partial Tumor Response by RECIST 1.0. Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: CT scan or MRI if used to follow lesion(s) for measurable disease every other cycle for the first 6 mnths; then every 3 mnths thereafter until dx progression is confirmed; also repeat any other time clinically indicated, assessed up to 6 months.
Population: Eligible and Treated Patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Pazopanib
Number analyzed (Participants) | 19
percentage of participants | 0 [0 to 14.6]

2. Primary Outcome: Percentage of Participants With Progression-free Survival (PFS) at 6 Months
Description: Progression-free survival is the period from study entry until disease progression, death or date of last contact. Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0), as a 20 % increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 6 months
Population: Eligible and treated patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Pazopanib
Number analyzed (Participants) | 19
percentage of participants | 15.8 [4.4 to 35.9]

3. Primary Outcome: Number of Patients With Grade 3 or Higher Adverse Events
Description: Grade 3 or higher adverse events were graded by CTCAE v4.
Time Frame: Every cycle while on treatment
Population: Eligible and Treated Patients
Measure: Number; unit: participants
Arm/Group | Pazopanib
Number analyzed (Participants) | 19
participants
  Anemia | 3
  Hypertension | 3
  Abdominal pain | 2
  Hyperglycemia | 2
  Hypoglycemia | 2
  Alanine aminotransferase increased | 1
  Ascites | 1
  Aspartate aminotransferase increased | 1
  Creatinine increasead | 1
  Death NOS | 1
  Dehydration | 1
  Diarrhea | 1
  Dyspnea | 1
  Fatigue | 1
  Headache | 1
  Hypocalcemia | 1
  Hyponatremia | 1
  Memory impairment | 1
  Nausea | 1
  Proctitis | 1
  Rectal hemorrhage | 1
  Sepsis | 1
  Vomiting | 1

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is the period from study entry until disease progression, death or date of last contact
Time Frame: From start of treatment to time of progression or death, assessed up to 5 years
Population: Eligible and Treated Patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pazopanib
Number analyzed (Participants) | 19
months | 2.0 [1.6 to 3.6]

5. Secondary Outcome: Overall Survival
Description: The observed length of life from entry into the study to death or the date of last contact.
Time Frame: Time from start of treatment to time of death or the date of last contact, assessed up to 5 years
Population: Eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pazopanib
Number analyzed (Participants) | 19
months | 8.7 [2.6 to 14.0]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported. Also reported are Serious Adverse Events (SAEs) for up to 5 years after stopping study treatment.
Arm/Group | Pazopanib
Serious Adverse Events (participants affected / at risk) | 6/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib (N=19)
Anemia (Blood and lymphatic system disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Death Nos (General disorders) | 1
Creatinine Increased (Investigations) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Memory Impairment (Nervous system disorders) | 1
Reproductive System And Breast Disorders - Other (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib (N=19)
Anemia (Blood and lymphatic system disorders) | 9
Sinus Bradycardia (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Hearing Impaired (Ear and labyrinth disorders) | 2
Ear Pain (Ear and labyrinth disorders) | 1
Blurred Vision (Eye disorders) | 3
Dysphagia (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 8
Bloating (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 7
Proctitis (Gastrointestinal disorders) | 1
Rectal Hemorrhage (Gastrointestinal disorders) | 2
Mucositis Oral (Gastrointestinal disorders) | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 1
Oral Pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 15
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Edema Trunk (General disorders) | 1
Edema Limbs (General disorders) | 1
Fatigue (General disorders) | 14
Fever (General disorders) | 1
Sinusitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Investigations - Other (Investigations) | 1
Weight Loss (Investigations) | 4
Platelet Count Decreased (Investigations) | 2
Lymphocyte Count Decreased (Investigations) | 1
Creatinine Increased (Investigations) | 2
Neutrophil Count Decreased (Investigations) | 10
Blood Bilirubin Increased (Investigations) | 3
White Blood Cell Decreased (Investigations) | 10
Aspartate Aminotransferase Increased (Investigations) | 4
Alkaline Phosphatase Increased (Investigations) | 3
Alanine Aminotransferase Increased (Investigations) | 4
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 6
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4
Neck Pain (Musculoskeletal and connective tissue disorders) | 2
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Peripheral Sensory Neuropathy (Nervous system disorders) | 8
Paresthesia (Nervous system disorders) | 1
Memory Impairment (Nervous system disorders) | 3
Headache (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 4
Anxiety (Psychiatric disorders) | 2
Urinary Retention (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 2
Pelvic Pain (Reproductive system and breast disorders) | 1
Vaginal Discharge (Reproductive system and breast disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 2
Nail Discoloration (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less